CLINICAL TRIAL: NCT05791747
Title: Representations, Beliefs and Attitudes Towards Hypnosis in Patients Followed for Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Nimes (Other)
Responsible Party: Principal Investigator, Baussard Louise, Associate professor, University of Nimes
Other Study IDs: UNimes3
Record Dates: First submitted 2023-03-14; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Cancer Colorectal; Hypnosis, Animal
Keywords: cancer colorectal; hypnose; representations
MeSH Terms: conditions — Colonic Neoplasms; Immobility Response, Tonic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: semi-structured interviews — This is an observational study Patients included in the study will conduct semi-structured interviews to discuss their knowledge and/or experience with supportive care, particularly hypnosis

SUMMARY:
Over the past decade, changes in knowledge and attitudes toward complementary and alternative medicine have been occurring. One study shows that 21% of patients are turning to them. In contrast, hypnosis is among the least used. While perceptions of alternative medicine are improving, there is still widespread skepticism about the beliefs of hypnosis and this may explain why patients are not turning to it. Although its use in oncology is no longer in question, and its efficacy in the management of side effects has been demonstrated, no recent qualitative study has been conducted to examine the representations of hypnosis among cancer patients. It therefore seems relevant to us today to know the evolution of the representations and attitudes of cancer patients towards hypnosis.

DETAILED DESCRIPTION:
Cancer patients experience psychological difficulties during the disease, associated with treatment, and even in the post-treatment period. Among the most common, they mention emotional distress, significant fatigue, sleep disturbance, or pain. Several authors agree that there is a cluster of four core symptoms associated with the disease and its treatments, including fatigue, nausea/vomiting, depression and pain. These symptoms have a significant impact on daily activities, resulting in a decrease in quality of life.

Reducing the symptoms of cancer to the sole etiology of the disease or its treatments does not allow us to consider a management action. Indeed, patients with cancer face the diagnosis and follow a course of care that includes many medical therapies (surgery, chemotherapy, radiotherapy, etc.). Integrative medicine takes into account the need for these medical therapies by adding the importance of supportive care for patients. Specifically, the expected effects are to reduce the after-effects for people thanks to an offer of support care adapted to their needs and regularly evaluated, ensuring a better quality of life immediately and in the longer term, as well as by providing information that allows patients to make the most informed choices possible.

Physical activity, dietary monitoring, and psychosocial interventions remain the most common complementary therapies offered to patients to reduce treatment side effects. Among this wide choice, patients can find themselves lost. Over the past decade, changes in knowledge and attitudes toward complementary and alternative medicine have been occurring. For example, one study found that 21% of patients are turning to them, indicating a growing interest in this type of care.

While perceptions of alternative medicine are improving, there is still widespread skepticism about hypnosis. As a result, even though scientific research shows positive effects of this type of therapy, a 2006 study in Canada found that out of 15 breast cancer patients using psychosocial therapies, only 6% used hypnosis. Another study conducted in 2018 confirms these results: on a population of 212 patients with different cancers, it appears that hypnosis is the therapy least used and whose interest is lowest.

Few studies have been conducted to determine the reasons for this lack of interest or the beliefs that are associated with hypnosis. Existing research suggests that patients lack information about hypnosis and its effectiveness, may have ambivalent perceptions about it or be skeptical of its effectiveness, and that their beliefs may be influenced by the media. Specifically, one study point out that positive attitudes toward hypnosis are even associated with better hypnotic response. While its use in oncology is no longer in question, no recent qualitative study has been conducted questioning the representations of hypnosis with cancer patients. It therefore seems relevant to us today to know the evolution of the representations and attitudes of cancer patients towards hypnosis. To do this, and according to Leventhal's model of self-regulation, the information obtained by a patient, whether or not it is medically based, is integrated by the patient in order to provide a "lay" understanding of the subject in question. Activated representations may then be guided by the individual's current and prior awareness or by social messages from perceived significant others or authoritative sources and this impacts attitudes.

The aim of the study was to investigate psychosocial representations related to hypnosis in colorectal cancer patients and to assess the impact of these representations on the intention to use hypnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Having been diagnosed with colorectal cancer
3. Able to understand and read French

Exclusion Criteria:

1. Patients who do not have a telephone or devices that allow remote interviewing
2. Medical (neurological, psychiatric, etc.) or psychological conditions that do not allow participation in the study (completion of the consent form and coherent speech for the interview)
3. Hearing impaired patient without hearing aids
4. Patient under guardianship or court protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women diagnosed with colorectal cancer, still in treatment or not.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-03-21 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
social representations | 30 minutes
  The representations will be questioned in terms of identity, beliefs, consequences, temporality and controlability. Semi-structured interviews with qualitative analyses will be conducted to explore represenations in cancer patients. The five major questions as are follows : What is hypnosis/hypnotherapy for you ? What do you think about hypnosis ? If you were to turn to this technique, what would be your expectations ? At what point in your illness/treatment would hypnosis be most appropriate ? Do you think hypnosis can help you manage the symptoms of your illness or the side effects of treatment ?

SECONDARY OUTCOMES:
Barriers and levers to using hypnosis | 30 minutes
  Identify what constitutes obstacles and levers to the use of hypnosis in analysing answers made at questions above
Intention to turn to hypnosis | 30 minutes
  What impacts intentions and attitudes towards hypnosis, semi-structured interviews will conclude with the following questions: - Do you intend to turn to this technique or refer a loved one ? What would make it easier for you to access hypnosis ?

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Nîmes, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: Yes
The principal investigator shares with the co-investigator the research protocol, consent, data collected
Supporting Information: Study Protocol, ICF
Time Frame: From january 2023 to december 2023 (one year)
Access Criteria: professionnal computer only

REFERENCES:
- [Background] Corbett, T., Groarke, A., Walsh, J. C., & McGuire, B. E. (2016). Cancer-related fatigue in post-treatment cancer survivors: Application of the common sense model of illness representations. BMC Cancer, 16(1), 919. https://doi.org/10.1186/s12885-016-2907-8 Curt, G. A., Breitbart, W., Cella, D., Groopman, J. E., Horning, S. J., Itri, L. M., Johnson, D. H., Miaskowski, C., Scherr, S. L., Portenoy, R. K., & Vogelzang, N. J. (2000). Impact of Cancer-Related Fatigue on the Lives of Patients: New Findings From the Fatigue Coalition. The Oncologist, 5(5), 353-360. https://doi.org/10.1634/theoncologist.5-5-353 Forlenza, M. J., Hall, P., Lichtenstein, P., Evengard, B., & Sullivan, P. F. (2005). Epidemiology of cancer-related fatigue in the Swedish twin registry. Cancer, 104(9), 2022-2031. Helyer, L. K., Chin, S., Chui, B. K., Fitzgerald, B., Verma, S., Rakovitch, E., Dranitsaris, G., & Clemons, M. (2006). The use of complementary and alternative medicines among patients with locally advanced breast cancer - a descriptive study. BMC Cancer, 6(1), 39. https://doi.org/10.1186/1471-2407-6-39 Henry, D. H., Viswanathan, H. N., Elkin, E. P., Traina, S., Wade, S., & Cella, D. (2008). Symptoms and treatment burden associated with cancer treatment: Results from a cross-sectional national survey in the U.S. Supportive Care in Cancer, 16(7), 791-801. https://doi.org/10.1007/s00520-007-0380-2 Hofman, M., Ryan, J. L., Figueroa-Moseley, C. D., Jean-Pierre, P., & Morrow, G. R. (2007). Cancer-Related Fatigue: The Scale of the Problem. The Oncologist, 12(S1), 4-10. https://doi.org/10.1634/theoncologist.12-S1-4 Lawrence, D. P. (2004). Evidence Report on the Occurrence, Assessment, and Treatment of Fatigue in Cancer Patients. Journal of the National Cancer Institute Monographs, 2004(32), 40-50. https://doi.org/10.1093/jncimonographs/lgh027 Leventhal, H., & Diefenbach, M. (1991). The Active Side of Illness Cognition. In J. A. Skelton & R. T. Croyle (Éds.), Mental Representation in Health and Illness (p. 247-272). Springer US. https://doi.org/10.1007/978-1-4613-9074-9_11 Lind, S. B., Jacobsen, H. B., Solbakken, O. A., & Reme, S. E. (2021). Clinical Hypnosis in Medical Care: A Mixed-Method Feasibility Study. Integrative Cancer Therapies, 20, 153473542110586. https://doi.org/10.1177/15347354211058678 Mendoza, M. E., Capafons, A., & Jensen, M. P. (2017). Hypnosis attitudes: Treatment effects and associations with symptoms in individuals with cancer. American Journal of Clinical Hypnosis, 60(1), 50-67. Miller, S. J., Schnur, J. B., Montgomery, G. H., & Jandorf, L. (2015). African-Americans and Latinos' Perceptions of Using Hypnosis to Alleviate Distress Before a Colonoscopy. NCCN. (2022). NCCN Clinical Practice Guidelines in Oncology-Cancer-Related Fatigue. NCCN.org. Qureshi, M., Zelinski, E., & Carlson, L. E. (2018). Cancer and Complementary Therapies: Current Trends in Survivors' Interest and Use. Integrative Cancer Therapies, 17(3), 844-853. https://doi.org/10.1177/1534735418762496